CLINICAL TRIAL: NCT03484039
Title: The Epilepsy Wellness Center: Incorporating Multidimensional Self-management Psychosocial Interventions in Epilepsy Care Improves the Well-being of Individuals With Epilepsy: a Feasibility and Proof-of-concept Study
Brief Title: Incorporating Multidimensional Psychosocial Interventions Improves the Well-being of Individuals With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Dupont Fund, Jesse Ball (Unknown); Florida Blue Foundation (Unknown); Riverside Hospital Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201800512
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy; Seizure Disorder
Keywords: memory problems; stress; depression; adherence; seizure documentation
MeSH Terms: conditions — Epilepsy; Memory Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in one module of own choice. Except for Module 3 Submodule 2, every module will consist of a particular intervention, as well as, its accompanying set of assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy Patients (Experimental): The group will receive the module (a 1-2 hour course on either medication adherence, seizure documentation, memory improvement or stress management) right after a baseline assessment. A post assessment and delayed post assessment will be conducted after the module is administered.
  Interventions: Behavioral: Medication Adherence; Behavioral: Seizure Documentation; Behavioral: Memory Improvement; Behavioral: Stress Management

INTERVENTIONS:
Behavioral: Medication Adherence — Some subjects will be enrolled in a medication adherence course.
Behavioral: Seizure Documentation — Some subjects will be enrolled in a seizure documentation course.
Behavioral: Memory Improvement — Some subjects will be enrolled in a memory improvement course.
Behavioral: Stress Management — Some subjects will be enrolled in a stress management course.

SUMMARY:
The purpose of this study is to incorporate multidimensional self-management programs into the routine care of epilepsy patients. Consenting patients will enroll in one of four interventions that help improve medication adherence, increase seizure awareness and documentation, improve memory and deal with stress and depression.

DETAILED DESCRIPTION:
Though tremendous advances have been made in the diagnosis and treatment of individuals with epilepsy, much remains to be done when it comes to improving their psychosocial well-being. Many individuals with epilepsy have difficulty adhering to treatment, documenting their seizure types, coping with memory difficulties, dealing with stress, and suffer from depression. These factors limit the quality of life of epilepsy patients and prevent them from realizing their full potential.

Patients will enroll in one of four interventions that help improve medication adherence, increase seizure awareness and documentation, improve memory and deal with stress and depression. Patient assessments will be conducted before and after intervention to gauge the efficacy of the programs.

The specific aims of this study are to assess the feasibility and patient acceptability of incorporating multidimensional self-management and psychosocial interventions into routine epileptic care, as well as, determine whether these incorporations improve self-management, quality-of-life, and other measures of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of epilepsy using established criteria
* Patient self-identified as own primary caregiver
* English fluency
* Ability to provide informed consent
* Ability to complete the study assessments

Exclusion Criteria:

* History of non-epileptic seizures
* History of cognitive impairments that prevents them from providing informed consent and completing study assessments

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life in Epilepsy-10 scores | To be administered at baseline (upon subject screening), pre-intervention (with 2 weeks prior to intervention), post-intervention (between 6 weeks to 3 months post-intervention), and delayed post-intervention (within 4&1/2 to 6 months post-intervention)
  This is a well-validated measure of quality of life for epilepsy patients. The unit of measure is a composite score ranging from 0-100 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Edmundo D Bautista, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided